CLINICAL TRIAL: NCT05677685
Title: Multicentre Randomized Double-blind Trial of VISUPRIME® Eye Drops to be Evaluated in Preventing the Conjunctival Bacterial Load in Patients Undergoing to Anti-VEGF Injection
Brief Title: VISUPRIME® Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VISUfarma SpA (Industry)
Collaborators: CROlife (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VF-03-2022
Record Dates: First submitted 2022-12-12; First posted 2023-01-10 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Macular Degeneration, Age Related; Myopic Choroidal Neovascularisation; Proliferative Diabetic Retinopathy; Diabetic Macular Edema; Macular Edema of Right Retina (Diagnosis)
MeSH Terms: conditions — Macular Degeneration; Disease

STUDY DESIGN:
Intervention Model Description: Eligible patients who meet the study inclusion criteria will be randomized in a 1:1 assignment ratio to the study group or control group in a double-blind manner.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study and therefore participants and clinical staff are not aware of the treatment group assigned to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Device (Active Comparator)
  Interventions: Device: VISUPRIME
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: VISUPRIME — twice daily
  Arms: Investigational Device
Device: Placebo — twice daily
  Arms: Placebo

SUMMARY:
The study purpose is to assess the efficacy of VISUPRIME® eye drops in preventing the conjunctival bacterial load in patients undergoing to anti-VEGF injection.

DETAILED DESCRIPTION:
Multicentre, double-masked, placebo-controlled randomized 1:1 of the VISUPRIME® treatment in patients undergoing intravitreal anti-VEGF injection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18)
* Naïve and pre-treated patients scheduled for IVI
* Diagnosis of one of the following:

  * ARMD
  * mCNV
  * Proliferative diabetic retinopathy
  * Diabetic macular oedema
  * Macular oedema secondary to retinal vein occlusion
* The subject has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, approved by the local Ethics Committee (EC).

Exclusion Criteria:

* Use of systemic antibiotics, corticosteroids within 3 months
* Use of topical antibiotics and or corticosteroids within 15 days from study enrolment
* Use of topical Artificial Tears within 15 days from the enrolment
* Use of topical antiseptic agents within 1 month from study enrolments
* Presence of topical ocular therapies that cannot be suspended for the entire duration of the study
* Ongoing ocular or systemic inflammatory or infectious processes
* Known hypersensitivity to the constituents of the study product
* Diagnosis of Open-Angle Glaucoma
* Uveitis
* Acute and Chronic Conjunctival Disease
* Any intraocular surgery within 6 months from study enrolment, excluded IVI
* Severe and Moderate Dry Eye
* Pregnancy or breast-feeding
* Participation in other clinical studies
* Patients with cognitive impairment and unable to manage home-assigned treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
CFU (Colony Forming Units) | three days
  Primary endpoint is to evaluate the change in bacterial loads in terms of CFU/ sample in the two groups at V0 compared to V1.

SECONDARY OUTCOMES:
Antibiotic sensitivity | three days
  Identification of microorganism sensitivity or resistant to various antibiotics using antibiogram technique.
SANDE Symptom Assessment iN Dry Eye | three days
  The assessment of ocular irritation symptoms at V0 and V1, using a 2-item Symptom Assessment iN Dry Eye (SANDE) questionnaire consistent with all ocular diseases that may impact vision-related functioning.
Adverse Events | three days
  Evaluation of the rate of related Adverse Events (AEs) that occur during the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rita Bigioni, PhD, Study Chair — CROlife
Locations (6):
- Italy (6):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, BA
  - Ospedale Santa Maria della Misericordia, Perugia, PG
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, RM
  - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste, TS
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara

IPD SHARING:
Plan to Share IPD: No